CLINICAL TRIAL: NCT04036721
Title: Randomized Open-label Study of the Impact of Prolonged Systemic Corticosteroid Therapy on the Course and Relapse Risk of Checkpoint Inhibitor Interstitial Lung Disease (Pneumonitis) Related to the Treatment of Solid Tumors With Anti-programmed-death Type 1 Receptor or Ligand Antibodies
Brief Title: Coorticosteroid Regimen in Patients With Anti-PD-1/PD-L1 Induced Pneumonitis
Acronym: PROS-CONS
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: SARS-CoV-2 cases stopped the recruitment in Organisation since July 2020
Sponsor: National Institute for Tuberculosis and Lung Diseases, Poland (Other)
Responsible Party: Principal Investigator, Mateusz Polaczek, Principal Investigator, National Institute for Tuberculosis and Lung Diseases, Poland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KB-57/2019
Record Dates: First submitted 2019-07-17; First posted 2019-07-30 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Lung Neoplasm Malignant; Interstitial Lung Disease
Keywords: anti-PD-1; anti-PD-L1; pneumonitis; NSCLC; treatment; programmed-death receptor
MeSH Terms: conditions — Lung Neoplasms; Lung Diseases, Interstitial; Pneumonia | interventions — Prednisone; Clinical Protocols

STUDY DESIGN:
Intervention Model Description: Randomization is 1:1 to Arms A and B, it will be conducted using adaptive minimization method. the randomization will be stratified upon three criteria:
  1. severity of suspected pneumonitis at baseline (G2 vs. G3-4)
  2. response for oncological treatment (PR and CR vs. SD and PD) 3) chronic respiratory system disorders The first patient will be randomized to Arm A or B with simple randomization method using computer program, this part will be oversight by medical monitor. The randomization will be performed for each patient by Primary Investigator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM A - PROLONGED (Experimental): induction dose 1-4mg/kg of prednisone, prednisone 60mg q24h for 2-4wks, tapering not faster than 10mg each 14d, maintenance dose 10mg q24h for 8wks, withdraw of treatment during 4wks, summary of treatment time not shorter than 12-24wks.
  Interventions: Drug: Prolonged glucocorticosteroid (prednisone) regimen
- ARM B - FAST REDUCTION (Active Comparator): induction dose 1-4mg/kg of prednisone, prednisone 30-60 mg q24h, tapering not faster than 10mg each 7d, summary of treatment time 6-12wks.
  Interventions: Drug: Short glucocorticosteroid (prednisone) regimen

INTERVENTIONS:
Drug: Prolonged glucocorticosteroid (prednisone) regimen — Prolongation of maintenance therapy with prednisone of patients with pneumonitis inducted by anyi-PD-1/anti-PD-L1 antibodies.
  Arms: ARM A - PROLONGED
Drug: Short glucocorticosteroid (prednisone) regimen — Prednison regimen based upon American Society of Clinical Oncology and European Society for Medical Oncology Clinical Practice Guidelines on pneumonitis treatment in patients receiving immunotherapy agents
  Arms: ARM B - FAST REDUCTION

SUMMARY:
This is a prospective interventional open-label randomized trial. The patients treated with anti-

PD-1 (programmed-death receptor type 1) or anti-PD-L1 (programmed-death ligand) antibodies in case of new acute onset interstitial changes or new seriuos respiratory system related symptoms will be recruited for this study to perform diagnostics. At the recruitment the patient will be randomized 1:1 to investigatory or control arm, the randomization will be stratified upon three criteria:

1. severity of suspected pneumonitis at baseline (grade 2 vs. grade 3-4)
2. response for oncological treatment (partial response (PR) and complete response (CR) vs. stable disease (SD) and progression disease (PD))
3. chronic respiratory system disorders Both groups will be treated in the same way in terms of diagnostic procedures. In case of interstitial lung diseases related to immune checkpoint inhibitor is confirmed with the severity of grade 2-4 in the modified CTCAE criteria the patient will get the treatment, accordingly to the randomization: ARM A - INVESTIGATORY GROUP the start dose will be 1-4 mg/kg of body weight of prednisone, depending on clinical condition and pneumonitis severity, the induction treatment will last for 5-7 days, in case of severe condition - no improvement after 48-72 h of initial treatment - introduction of immunosuppressive agent is recommended - cyclophosphamide, mofetil mycophenolate or infliximab. A continuation treatment with dose tapering is than recommended, starting from 60mg q 24h of prednisone for 2-4 weeks, and dropping the dose 10mg q 24 h not faster than over 14 days; the maintenance dose of prednisone 10mg q 24 h should be hold for 8 weeks and withdraw should last for 4 weeks. This arm will be treated with corticosteroid for at least 12-24 weeks.

ARM B - CONTROL GROUP the starting dose will be 1-4mg/kg of body weight of prednisone , depending on clinical condition and pneumonitis severity, the induction treatment will last 5-7 days; in case of severe condition - no improvement after 48-72 h of initial treatment - introduction of immunosuppressive agent is recommended: cyclophosphamide, mofetil mycophenolate or infliximab. A continuation treatment with dose tapering is than planned, starting from oral dose of 30-60mg q 24h of prednisone, and dose reduction of 10mg q 24 h each 1 week. This arm will be treated for 6-12 weeks.

During the treatment and after its termination the function of respiratory system, interstitial changes in radiologic examinations, anticancer response, survival time, pneumonitis relapse and glucocorticosteroid side effects will be monitored and evaluated. The observation will last up to 52 weeks.

DETAILED DESCRIPTION:
1. Diagnostic period The screening for the study will involve patients with newly diagnosed interstitial changes in chest radiological examination or in patient with new respiratory system related symptoms. The radiological changes must be confirmed in chest computed tomography (CT). In case on inclusion criteria are meet the patient will be randomized and will begin the diagnostic process.

In both groups the diagnostic process will be the same, based upon the existing recommendations it will involve:

1. detailed medical history and physical examination;
2. laboratory tests: CBC, CRP, PCT, ALT, AST, CK, LDH, Na, K, Ca, glucose, proteinogram, flow cytometry, IgG and IgM levels, anti-nuclear antibodies (immunofluorescence, dilution), cytomegalovirus (CMV) polymerase-chain reaction (PCR), IgG and IgM for Legionella pneumophila, Chlamydia pneumoniae, Mycoplasma pneumoniae, QuantiferonTB-GOLD, NT- proBNP, troponin T;
3. arterialized blood gas panel;
4. in case it was not yet performed - chest computed tomography with contras enhancement with exclusion of pulmonary embolism;
5. 12-lead electrocardiograph
6. spirometry, full body plethysmography with carbon monoxide diffusion, 6-minute walk test
7. flexible bronchoscopy with:

   1. culture for aerobic bacteria
   2. culture for Mycobacterium tuberculosis (TB), TB PCR,
   3. culture for funguses, Aspergillus antigen, PCR and immunofluoroscopic examination for Pneumocystis jiroveci (PCP)
   4. bronchoalveolar lavage (BAL) with BAL fluid cell analysis
   5. transbronchial lung biopsy with forceps or nitrogen-criobiopsy, exclusion of CMV pneumonia and neoplasm progression, histological examination for pneumonitis histological pattern; bronchoalveolar lavage and lung biopsy will be performed only in patient with no clinical contradictions.

      Interstitial lung diseases related to immune checkpoint inhibitor, i.e. interstitial pneumonia related to checkpoint inhibitor or immunotherapy, i.e. pneumonitis: definition:

      the appearance of new radiological changes in chest examination (chest CT or plain radiogram proved with chest CT) after being exposed (treated) with anti-PD-1 or anti-PD-L1 monoclonal antibody, the radiological changes can be described as interstitial: ground glass opacities, consolidations with air bronchogram, interstitial septa thickening, central lobular nodules with perilymphatic distribution; the changes cannot be explained with neoplasm progression, active respiratory infection, heart failure or one of the above is not a sole explanation for the changes. The radiological changes are sometimes accompanied with respiratory system related symptoms. Each case need detailed differential and diagnosis of pneumonitis diagnosis can be made established after active exclusion of other potential causes. Good reaction for glucocorticosteroid treatment makes the diagnosis more likely.

      The severity of pneumonitis should be based on 5 point scale based on the modified Common Terminology for Adverse Events (CTC AE) v. 5 criteria:

      Grade 1 (G1) Interstitial changes with no symptoms and no progression in follow-up examination after few days.

      Grade 2 (G2) Interstitial changes without respiratory failure with mild to moderate respiratory symptoms.

      Each case of asymptomatic relapse. Grade 3 (G3) Interstitial changes with acute respiratory failure and the need of oxygen therapy.

      Grade 4 (G4) Interstitial changes with acute respiratory failure and the need of mechanical ventilation.

      Grade 5 (G5) Death related to acute interstitial pneumonitis.

      The diagnostics and treatment of patient should be based on patients condition and conducted in pulmonology or intensive care unit (ICU) department. The treatment should always be driven by the most likely diagnosis and the participation in the study should not delay any procedure or medication administration.

      In cases when radiological changes were discovered and severity is grade 1 it is recommended to perform a follow up chest radiograph after 5-7 days to see the dynamics and reassess the severity.

      2. Induction treatment General rules: The treatment is conducted based on patients condition in ICU or pulmonology department. The commence of glucocorticosteroid administration should take place with no delay in patient with high suspicion of grade 4 pneumonitis (max. 12 h after the beginning of diagnostics), in case of grade 3 pneumonitis the time to the initiation of treatment should last less than 24 h, and in grade 2 pneumonitis the diagnostics should last no longer than 5 days. The induction treatment last for 5-7 days.

      In case of elevated inflammatory markers, clinical, laboratory or microbiological signs of infection accompanying pneumonitis it is recommended to administer antibiotics. Antibiotics will not be routinely used in the whole study population.

      Arm A: initial dose in grade 2 is 1 mg/kg of body weight of oral prednisone, in grade 3-4 - 2- 4mg/kg of body weight of intravenous methylprednisolone, depending on severity and clinical condition. Induction treatment for 5-7 days; in cases of severe course - bad condition and no improvement after initial 48-72 h - introduction of cyclophosphamide, mycophenolate mofetile or infliximab.

      Arm B: initial dose in grade 2 is 1 mg/kg of body weight of oral prednisone, in grade 3-4 - 2- 4mg/kg of body weight of intravenous methylprednisolone, depending on severity and clinical condition. Induction treatment for 5-7 days; in cases of severe course - bad condition and no improvement after initial 48-72 h - introduction of cyclophosphamide, mycophenolate mofetile or infliximab.

      Dosage and administration: Preferred intravenous corticosteroid is methylprednisolone, the dosage range is 1-4 mg/kg of body weight, but in case 4mg/kg is considered a flat dose of 500mg q 24 h is recommended. The medication will be diluted in saline, it will be administered in single daily dose.

      The preferred oral medication is prednisone, dosage is 1mg/kg of body weight, but not more than 60mg, administered in single dose daily.

      The administration of cyclophosphamide, mycophenolate mofetile or infliximab will be based on case-by-case decision of multidisciplinary board and dosage will be based on the summary of the medical product characteristics.

      3. Maintenance treatment General rules: the treatment should start the last day of induction treatment if intravenous corticosteroid was administered, in case of oral induction treatment it should start the next day after induction in over. It is based on oral medication, administered in one daily dose in the morning. In case of grade 2 pneumonitis the immunotherapy re-challenge is possible after the dose of 10mg q 24h of prednisone is reached. The dose modification should be considered in case of serious side effects of steroid therapy.

      During glucocorticosteroid therapy no routine prophylaxis of pneumocystis pneumonia is recommended, and the administration of co-trimoxazole should be analyzed case by case; it should be considered in cases of positive PCR results for Pneumocystis jiroveci and in patient with T C4+ cells depletion in flow cytometry - less than 200 cells per microliter. During steroid therapy osteoporosis prophylaxis can be considered. We do not recommend antifungal prophylaxis.

      Arm A: The maintenance treatment with oral agent, the general rules must be meet - tapering starts at the dose of 60mg q 24 h of prednisone for 2-4 weeks, the reduction is not faster than 10mg each 14 days, the maintenance dose if flat 10mg q 24 h dose for 8 weeks and the withdraw should be slow over 4 weeks. The treatment should last 12-24 weeks or longer. The detailed dose of daily prednisone is presented in Tables.

      Arm B: Treatment with oral agent, based on general rules - the tapering starts at the dose of 30- 60 mg q 24h of prednisone, the reduction is no faster than 10mg each 7 days, the treatment lasts between 6 and 12 weeks. The detailed dosage proposition is presented in the Tables.

      Dosage and administration: The preferred oral agent is prednisone, in single daily dose administered in the morning. The recommended dose of co-trimoxazole in case of PCP prophylaxis is 960mg q2d administered on Monday, Wednesday and Friday; it should last until 10mg q 24h of prednisone is reached.

      4. Relapse treatment In case of relapse suspicion the workup should be the same as initial starting from the diagnostic period. The treatment scheme is as in Arm A.

      5. Follow-up period The observation starts from the first day of the maintenance therapy. The clinical and radiological follow-up is planned each 4-6 weeks during the first 24 weeks and then each 12 weeks. The observation will last up to 52 weeks. In the follow-up points steroid side effects, anticancer response, treatment efficacy and signs of relapse will be evaluated, using:

1) detailed history and physical examination 2) chest radiogram

In the 12 weeks (t12) and 52 weeks (t52) point follow-up extra procedures to exaluate the endpoint will be performed:

1. chest computed tomography
2. arterialized blood gas panel
3. spirometry, full body plethysmography with carbon monoxide diffusion, 6-minute walk test

ELIGIBILITY:
Inclusion Criteria:

1. age over 18 years old
2. histological or cytological confirmation of solid cancer
3. treatment with anti-PD-1 or anti-PD-L1 antibody in monotherapy or in combination with cytotoxic chemotherapy or antiangiogenic agents like anti-vascular epitheliar growth factor antibodies
4. acute onset respiratory symptoms or lung changes in radiologic examinations which were not present before immunotherapy was introduced e. signed informed consent

Exclusion Criteria:

1. concomitant or previous treatment with anti-CTLA4 or other immunotherapeutic agents
2. active untreated tuberculosis
3. the use of glucocorticosteroids in the dose equivalent to 10mg q 24h or more of prednisone in the last 4 weeks in indication other than pneumonitis or different immune related adverse event d. withdraw of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Pneumonitis relapse | 12 months
  Incidence of pneumonitis relapse in study arm A vs. control arm B
Pneumonitis related deaths | 12 months
  Incidence of pneumonitis related deaths in arm A vs. arm B
Radiological regression of pneumonitis | 12 weeks and 52 weeks
  Computed tomography assesment of pneumonitis regression, compared to initial examination. 4-point scale: coplete regression, definite partial response, slight partial response, progression.

SECONDARY OUTCOMES:
Overall survival | 12 months
  Overall survival in study arm vs. control arm - incidence of deaths in arm A vs. arm B
Progression-free survival | 12 months
  Progression-free survival in study arm vs. control arm - no clinical or radiological signs of neoplasm progression
Incidence of treatment related adverse events. | 12 months
  Corticosteroid related side effects - event or serious adverse event (need for faster dose reduction or additional treatment).

OTHER OUTCOMES:
Diagnostic procedure evaluation | 1 week
  Number of certain cases and number of uncertain cases in terms of pneumonitis diagnosis will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Instutut Gruzlicy I Chorob Pluc, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rittmeyer A, Barlesi F, Waterkamp D, Park K, Ciardiello F, von Pawel J, Gadgeel SM, Hida T, Kowalski DM, Dols MC, Cortinovis DL, Leach J, Polikoff J, Barrios C, Kabbinavar F, Frontera OA, De Marinis F, Turna H, Lee JS, Ballinger M, Kowanetz M, He P, Chen DS, Sandler A, Gandara DR; OAK Study Group. Atezolizumab versus docetaxel in patients with previously treated non-small-cell lung cancer (OAK): a phase 3, open-label, multicentre randomised controlled trial. Lancet. 2017 Jan 21;389(10066):255-265. doi: 10.1016/S0140-6736(16)32517-X. Epub 2016 Dec 13. PMID 27979383
- [Background] Socinski MA, Jotte RM, Cappuzzo F, Orlandi F, Stroyakovskiy D, Nogami N, Rodriguez-Abreu D, Moro-Sibilot D, Thomas CA, Barlesi F, Finley G, Kelsch C, Lee A, Coleman S, Deng Y, Shen Y, Kowanetz M, Lopez-Chavez A, Sandler A, Reck M; IMpower150 Study Group. Atezolizumab for First-Line Treatment of Metastatic Nonsquamous NSCLC. N Engl J Med. 2018 Jun 14;378(24):2288-2301. doi: 10.1056/NEJMoa1716948. Epub 2018 Jun 4. PMID 29863955
- [Background] Borghaei H, Paz-Ares L, Horn L, Spigel DR, Steins M, Ready NE, Chow LQ, Vokes EE, Felip E, Holgado E, Barlesi F, Kohlhaufl M, Arrieta O, Burgio MA, Fayette J, Lena H, Poddubskaya E, Gerber DE, Gettinger SN, Rudin CM, Rizvi N, Crino L, Blumenschein GR Jr, Antonia SJ, Dorange C, Harbison CT, Graf Finckenstein F, Brahmer JR. Nivolumab versus Docetaxel in Advanced Nonsquamous Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Oct 22;373(17):1627-39. doi: 10.1056/NEJMoa1507643. Epub 2015 Sep 27. PMID 26412456
- [Background] Gandhi L, Rodriguez-Abreu D, Gadgeel S, Esteban E, Felip E, De Angelis F, Domine M, Clingan P, Hochmair MJ, Powell SF, Cheng SY, Bischoff HG, Peled N, Grossi F, Jennens RR, Reck M, Hui R, Garon EB, Boyer M, Rubio-Viqueira B, Novello S, Kurata T, Gray JE, Vida J, Wei Z, Yang J, Raftopoulos H, Pietanza MC, Garassino MC; KEYNOTE-189 Investigators. Pembrolizumab plus Chemotherapy in Metastatic Non-Small-Cell Lung Cancer. N Engl J Med. 2018 May 31;378(22):2078-2092. doi: 10.1056/NEJMoa1801005. Epub 2018 Apr 16. PMID 29658856
- [Background] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Yokoi T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Wadsworth C, Melillo G, Jiang H, Huang Y, Dennis PA, Ozguroglu M; PACIFIC Investigators. Durvalumab after Chemoradiotherapy in Stage III Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Nov 16;377(20):1919-1929. doi: 10.1056/NEJMoa1709937. Epub 2017 Sep 8. PMID 28885881
- [Background] Travis WD, Costabel U, Hansell DM, King TE Jr, Lynch DA, Nicholson AG, Ryerson CJ, Ryu JH, Selman M, Wells AU, Behr J, Bouros D, Brown KK, Colby TV, Collard HR, Cordeiro CR, Cottin V, Crestani B, Drent M, Dudden RF, Egan J, Flaherty K, Hogaboam C, Inoue Y, Johkoh T, Kim DS, Kitaichi M, Loyd J, Martinez FJ, Myers J, Protzko S, Raghu G, Richeldi L, Sverzellati N, Swigris J, Valeyre D; ATS/ERS Committee on Idiopathic Interstitial Pneumonias. An official American Thoracic Society/European Respiratory Society statement: Update of the international multidisciplinary classification of the idiopathic interstitial pneumonias. Am J Respir Crit Care Med. 2013 Sep 15;188(6):733-48. doi: 10.1164/rccm.201308-1483ST. PMID 24032382
- [Background] Suresh K, Voong KR, Shankar B, Forde PM, Ettinger DS, Marrone KA, Kelly RJ, Hann CL, Levy B, Feliciano JL, Brahmer JR, Feller-Kopman D, Lerner AD, Lee H, Yarmus L, D'Alessio F, Hales RK, Lin CT, Psoter KJ, Danoff SK, Naidoo J. Pneumonitis in Non-Small Cell Lung Cancer Patients Receiving Immune Checkpoint Immunotherapy: Incidence and Risk Factors. J Thorac Oncol. 2018 Dec;13(12):1930-1939. doi: 10.1016/j.jtho.2018.08.2035. Epub 2018 Sep 26. PMID 30267842
- [Background] Haanen JBAG, Carbonnel F, Robert C, Kerr KM, Peters S, Larkin J, Jordan K; ESMO Guidelines Committee. Management of toxicities from immunotherapy: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2018 Oct 1;29(Suppl 4):iv264-iv266. doi: 10.1093/annonc/mdy162. No abstract available. PMID 29917046
- [Background] Brahmer JR, Lacchetti C, Schneider BJ, Atkins MB, Brassil KJ, Caterino JM, Chau I, Ernstoff MS, Gardner JM, Ginex P, Hallmeyer S, Holter Chakrabarty J, Leighl NB, Mammen JS, McDermott DF, Naing A, Nastoupil LJ, Phillips T, Porter LD, Puzanov I, Reichner CA, Santomasso BD, Seigel C, Spira A, Suarez-Almazor ME, Wang Y, Weber JS, Wolchok JD, Thompson JA; National Comprehensive Cancer Network. Management of Immune-Related Adverse Events in Patients Treated With Immune Checkpoint Inhibitor Therapy: American Society of Clinical Oncology Clinical Practice Guideline. J Clin Oncol. 2018 Jun 10;36(17):1714-1768. doi: 10.1200/JCO.2017.77.6385. Epub 2018 Feb 14. PMID 29442540
- [Background] Delaunay M, Cadranel J, Lusque A, Meyer N, Gounant V, Moro-Sibilot D, Michot JM, Raimbourg J, Girard N, Guisier F, Planchard D, Metivier AC, Tomasini P, Dansin E, Perol M, Campana M, Gautschi O, Fruh M, Fumet JD, Audigier-Valette C, Couraud S, Dalle S, Leccia MT, Jaffro M, Collot S, Prevot G, Milia J, Mazieres J. Immune-checkpoint inhibitors associated with interstitial lung disease in cancer patients. Eur Respir J. 2017 Aug 10;50(2):1700050. doi: 10.1183/13993003.00050-2017. Print 2017 Aug. PMID 28798088
- [Background] Naidoo J, Wang X, Woo KM, Iyriboz T, Halpenny D, Cunningham J, Chaft JE, Segal NH, Callahan MK, Lesokhin AM, Rosenberg J, Voss MH, Rudin CM, Rizvi H, Hou X, Rodriguez K, Albano M, Gordon RA, Leduc C, Rekhtman N, Harris B, Menzies AM, Guminski AD, Carlino MS, Kong BY, Wolchok JD, Postow MA, Long GV, Hellmann MD. Pneumonitis in Patients Treated With Anti-Programmed Death-1/Programmed Death Ligand 1 Therapy. J Clin Oncol. 2017 Mar;35(7):709-717. doi: 10.1200/JCO.2016.68.2005. Epub 2016 Sep 30. PMID 27646942
- [Background] Cordier JF. Cryptogenic organising pneumonia. Eur Respir J. 2006 Aug;28(2):422-46. doi: 10.1183/09031936.06.00013505. PMID 16880372
- [Background] Suresh K, Naidoo J, Lin CT, Danoff S. Immune Checkpoint Immunotherapy for Non-Small Cell Lung Cancer: Benefits and Pulmonary Toxicities. Chest. 2018 Dec;154(6):1416-1423. doi: 10.1016/j.chest.2018.08.1048. Epub 2018 Sep 4. PMID 30189190